CLINICAL TRIAL: NCT02247349
Title: A Phase 1/2 Multicenter Study of BMS-986012 in Subjects With Relapsed/Refractory Small Cell Lung Cancer
Brief Title: BMS-986012 in Relapsed/Refractory SCLC
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CA001-030; 2014-002372-89 (EudraCT Number)
Record Dates: First submitted 2014-09-19; First posted 2014-09-25 (Estimated); Results first posted 2024-03-05 (Actual); Last update posted 2024-03-05 (Actual); Status verified 2024-02

CONDITIONS: Small Cell Lung Cancer
MeSH Terms: conditions — Small Cell Lung Carcinoma | interventions — Nivolumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (12):
- Dose Escalation (Monotherapy) Dose -1 (Experimental): BMS-986012 (anti-fucosyl-GM1) Intravenous solution once every 3 weeks until disease progression/clinical deterioration or unacceptable toxicity
  Interventions: Biological: BMS-986012 (anti-fucosyl-GM1)
- Dose Escalation (Monotherapy) Dose 1 (Experimental): BMS-986012 (anti-fucosyl-GM1) Intravenous solution once every 3 weeks until disease progression/clinical deterioration or unacceptable toxicity
  Interventions: Biological: BMS-986012 (anti-fucosyl-GM1)
- Dose Escalation (Monotherapy) Dose 2 (Experimental): BMS-986012 (anti-fucosyl-GM1) Intravenous solution once every 3 weeks until disease progression/clinical deterioration or unacceptable toxicity
  Interventions: Biological: BMS-986012 (anti-fucosyl-GM1)
- Dose Escalation (Monotherapy) Dose 3 (Experimental): BMS-986012 (anti-fucosyl-GM1) Intravenous solution once every 3 weeks until disease progression/clinical deterioration or unacceptable toxicity
  Interventions: Biological: BMS-986012 (anti-fucosyl-GM1)
- Dose Escalation (Monotherapy) Dose 4 (Experimental): BMS-986012 (anti-fucosyl-GM1) Intravenous solution once every 3 weeks until disease progression/clinical deterioration or unacceptable toxicity
  Interventions: Biological: BMS-986012 (anti-fucosyl-GM1)
- Dose Expansion (Monotherapy)- Cohort A (Refractory) (Experimental): BMS-986012 (anti-fucosyl-GM1) Intravenous solution once every 3 weeks until disease progression/clinical deterioration or unacceptable toxicity
  Interventions: Biological: BMS-986012 (anti-fucosyl-GM1)
- Dose Expansion (Monotherapy) Cohort B (Refractory) (Experimental): BMS-986012 (anti-fucosyl-GM1) Intravenous solution once every 3 weeks until disease progression/clinical deterioration or unacceptable toxicity
  Interventions: Biological: BMS-986012 (anti-fucosyl-GM1)
- Dose Expansion (Monotherapy) Cohort C (Sensitive) (Experimental): BMS-986012 (anti-fucosyl-GM1) Intravenous solution once every 3 weeks until disease progression/clinical deterioration or unacceptable toxicity
  Interventions: Biological: BMS-986012 (anti-fucosyl-GM1)
- Dose Expansion (Monotherapy) Cohort D (Sensitive) (Experimental): BMS-986012 (anti-fucosyl-GM1) Intravenous solution once every 3 weeks until disease progression/clinical deterioration or unacceptable toxicity
  Interventions: Biological: BMS-986012 (anti-fucosyl-GM1)
- Dose Escalation (Combination) Dose 1 (Experimental): BMS-986012 (anti-fucosyl-GM1) Intravenous solution once every 3 weeks until disease progression/clinical deterioration or unacceptable toxicity in combination with Nivolumab specified dose on specified days
  Interventions: Biological: BMS-986012 (anti-fucosyl-GM1); Biological: Nivolumab
- Dose Escalation (Combination) Dose 2 (Experimental): BMS-986012 (anti-fucosyl-GM1) Intravenous solution once every 3 weeks until disease progression/clinical deterioration or unacceptable toxicity in combination with Nivolumab specified dose on specified days
  Interventions: Biological: BMS-986012 (anti-fucosyl-GM1); Biological: Nivolumab
- Dose Expansion (Combination)- (Refractory and Sensitive) (Experimental): BMS-986012 (anti-fucosyl-GM1) Intravenous solution once every 3 weeks until disease progression/clinical deterioration or unacceptable toxicity in combination with Nivolumab specified dose on specified days
  Interventions: Biological: BMS-986012 (anti-fucosyl-GM1); Biological: Nivolumab

INTERVENTIONS:
Biological: BMS-986012 (anti-fucosyl-GM1)
Biological: Nivolumab
  Arms: Dose Escalation (Combination) Dose 1; Dose Escalation (Combination) Dose 2; Dose Expansion (Combination)- (Refractory and Sensitive)

SUMMARY:
The purpose of this study is to determine the safety, tolerability, pharmacokinetics, immunogenicity, antitumor activity and pharmacodynamics of BMS-986012 alone and in combination with nivolumab in patients with relapsed/refractory SCLC.

ELIGIBILITY:
For more information regarding BMS clinical trial participation, please visit www.BMSStudyConnect.com

Inclusion Criteria:

* Histological or cytological confirmed small cell lung cancer (SCLC)
* Performance Status 0-1
* Adequate organ function
* Measurable disease

Exclusion Criteria:

* Known or suspected brain metastasis
* Small cell cancer not lung in origin
* Significant or acute medical illness
* Uncontrolled or significant cardiac disease
* Infection
* ≥ Grade 2 peripheral neuropathy
* Concomitant malignancies
* HIV related disease or known or suspected HIV+
* Hepatitis B or C infection
* ECG abnormalities as defined by the protocol
* Allergies or hypersensitivities to monoclonal antibodies, BMS-986012 or related compounds, including fucosyl-GM1 vaccine and Nivolumab

Other protocol defined inclusion/exclusion criteria could apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 106 (Actual)
Dates: Start 2014-11-14 (Actual); Primary Completion 2022-12-21 (Actual); Study Completion 2022-12-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (16):
- United States (3):
  - Local Institution - 0004, New York, New York
  - Local Institution - 0001, Durham, North Carolina
  - Local Institution - 0021, Winston-Salem, North Carolina
- Australia (3):
  - Local Institution - 0020, St Leonards, New South Wales
  - Local Institution - 0011, Brisbane, Queensland
  - Local Institution - 0002, Clayton, Victoria
- Belgium (2):
  - Local Institution - 0015, Ghent
  - Local Institution - 0012, Liège
- Canada (5):
  - Local Institution - 0003, Edmonton, Alberta
  - Local Institution - 0017, Halifax, Nova Scotia
  - Local Institution - 0019, Hamilton, Ontario
  - Local Institution - 0010, London, Ontario
  - Local Institution - 0007, Toronto, Ontario
- Local Institution - 0013, Nijmegen, Netherlands
- Local Institution - 0009, San Juan, Puerto Rico
- Local Institution - 0008, Seoul, South Korea

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: FDA Safety Alerts and Recalls — http://www.fda.gov/safety/medwatch/safetyinformation/default.htm
- See also: BMS Clinical Trial Patient Recruiting — http://www.BMSStudyConnect.com
- See also: Related Info — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217331&parentIdentifier=CA001-030&attachmentIdentifier=938d9963-10f4-416b-94f0-d0b0f2d32930&fileName=ca001030-protamend03-redacted-final-.pdf&versionIdentifier=

RESULTS

PARTICIPANT FLOW:
Groups:
- BMS 70mg: 70 mg IV BMS-986012 every 21 days until protocol-specified discontinuation criteria are met
- BMS 160mg: 160 mg IV BMS-986012 every 21 days until protocol-specified discontinuation criteria are met
- BMS 400mg: 400 mg IV BMS-986012 every 21 days until protocol-specified discontinuation criteria are met
- BMS 1000mg: 1000 mg IV BMS-986012 every 21 days until protocol-specified discontinuation criteria are met
- BMS 400mg + Nivo 360mg: 400 mg IV BMS-986012 + 360 mg Nivolumab every 21 days until protocol-specified discontinuation criteria are met
- BMS 1000mg + Nivo 360mg: 1000 mg IV BMS-986012 + 360 mg Nivolumab every 21 days until protocol-specified discontinuation criteria are met
Period: Overall Study
Arm/Group | BMS 70mg | BMS 160mg | BMS 400mg | BMS 1000mg | BMS 400mg + Nivo 360mg | BMS 1000mg + Nivo 360mg
Started | 7 | 6 | 29 | 35 | 21 | 8
Completed | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 7 | 6 | 29 | 35 | 21 | 8
Not completed — Disease Progression | 7 | 4 | 26 | 31 | 16 | 6
Not completed — Study drug toxicity | 0 | 1 | 1 | 1 | 2 | 2
Not completed — Death | 0 | 0 | 0 | 1 | 0 | 0
Not completed — Adverse Event unrelated to study drug | 0 | 0 | 0 | 0 | 1 | 0
Not completed — Participant request to discontinue study treatment | 0 | 0 | 1 | 2 | 1 | 0
Not completed — Withdrawal by Subject | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Administrative reason by sponsor | 0 | 0 | 0 | 0 | 1 | 0
Not completed — Other reasons | 0 | 0 | 1 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | BMS 70mg | BMS 160mg | BMS 400mg | BMS 1000mg | BMS 400mg + Nivo 360mg | BMS 1000mg + Nivo 360mg | Total
Number analyzed (Participants) | 7 | 6 | 29 | 35 | 21 | 8 | 106
Age, Continuous [Mean (Standard Deviation); unit: Years] | 65.1 (10.6) | 58.3 (8.1) | 64.4 (9.2) | 61.7 (9.5) | 62.1 (9.8) | 61.1 (7.3) | 62.5 (9.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 4 | 11 | 12 | 9 | 5 | 45
  Male | 3 | 2 | 18 | 23 | 12 | 3 | 61
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 1 | 0 | 1 | 0 | 3
  Not Hispanic or Latino | 6 | 6 | 26 | 33 | 20 | 8 | 99
  Unknown or Not Reported | 0 | 0 | 2 | 2 | 0 | 0 | 4
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 1 | 3 | 0 | 0 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 1 | 0 | 0 | 0 | 1
  White | 7 | 6 | 27 | 30 | 21 | 8 | 99
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 2 | 0 | 0 | 2

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Events (AEs)
Description: Number of participants with any grade adverse events (AEs). An Adverse Event (AE) is defined as any new untoward medical occurrence or worsening of a pre-existing medical condition in a clinical investigation participant administered study drug and that does not necessarily have a causal relationship with this treatment. Toxicities will be graded using the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version 4.03.
Time Frame: From first dose to 100 days post last dose (Up to 64 months)
Population: All treated participants
Measure: Count of Participants; unit: Participants
Arm/Group | BMS 70mg | BMS 160mg | BMS 400mg | BMS 1000mg | BMS 400mg + Nivo 360mg | BMS 1000mg + Nivo 360mg
Number analyzed (Participants) | 7 | 6 | 29 | 35 | 21 | 8
Participants | 7 | 6 | 29 | 35 | 21 | 8

2. Primary Outcome: Number of Participants With Serious Adverse Events (SAEs)
Description: Number of participants with any grade serious adverse events (SAEs). A Serious Adverse Event (SAE) is any untoward medical occurrence that at any dose:
  * results in death
  * is life-threatening
  * requires inpatient hospitalization or causes prolongation of existing hospitalization
  * results in persistent or significant disability/incapacity
  * is a congenital anomaly/birth defect
  * is an important medical event Toxicities will be graded using the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version 4.03.
Time Frame: From first dose to 100 days post last dose (Up to 64 months)
Population: All treated participants
Measure: Count of Participants; unit: Participants
Arm/Group | BMS 70mg | BMS 160mg | BMS 400mg | BMS 1000mg | BMS 400mg + Nivo 360mg | BMS 1000mg + Nivo 360mg
Number analyzed (Participants) | 7 | 6 | 29 | 35 | 21 | 8
Participants | 7 | 4 | 21 | 24 | 11 | 5

3. Primary Outcome: Number of Participants With Adverse Events (AEs) Leading to Discontinuation
Description: Number of participants with any grade adverse events (AEs) leading to discontinuation. An Adverse Event (AE) is defined as any new untoward medical occurrence or worsening of a pre-existing medical condition in a clinical investigation participant administered study drug and that does not necessarily have a causal relationship with this treatment. Toxicities will be graded using the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version 4.03.
Time Frame: From first dose to 100 days post last dose (Up to 64 months)
Population: All treated participants
Measure: Count of Participants; unit: Participants
Arm/Group | BMS 70mg | BMS 160mg | BMS 400mg | BMS 1000mg | BMS 400mg + Nivo 360mg | BMS 1000mg + Nivo 360mg
Number analyzed (Participants) | 7 | 6 | 29 | 35 | 21 | 8
Participants | 0 | 1 | 2 | 5 | 3 | 2

4. Primary Outcome: Number of Participants Who Died
Description: Number of participants who died due to any cause.
Time Frame: From first dose to 100 days post last dose (Up to 64 months)
Population: All treated participants
Measure: Count of Participants; unit: Participants
Arm/Group | BMS 70mg | BMS 160mg | BMS 400mg | BMS 1000mg | BMS 400mg + Nivo 360mg | BMS 1000mg + Nivo 360mg
Number analyzed (Participants) | 7 | 6 | 29 | 35 | 21 | 8
Participants | 3 | 2 | 10 | 16 | 2 | 4

5. Primary Outcome: Number of Participants With Abnormal Hepatic Test
Description: Number of participants with laboratory abnormalities in specific hepatic tests. The number of participants with the following laboratory abnormalities from on-treatment evaluations will be summarized:
  * ALT or AST > 5xULN, > 3xULN, and > 2xULN
  * Any of ALT, AST, Total Bilirubin or ALP > 8xULN
  * Total bilirubin > 3xULN
  ALT = Alanine Aminotransferase; AST = Aspartate Aminotransferase; ULN = Upper Limit of Normal
Time Frame: From first dose to 100 days post last dose (Up to 64 months)
Population: All treated participants
Measure: Count of Participants; unit: Participants
Arm/Group | BMS 70mg | BMS 160mg | BMS 400mg | BMS 1000mg | BMS 400mg + Nivo 360mg | BMS 1000mg + Nivo 360mg
Number analyzed (Participants) | 7 | 6 | 29 | 35 | 21 | 8
Participants
  ALT OR AST > 5XULN | 0 | 0 | 0 | 1 | 1 | 2
  ALT OR AST > 3XULN | 0 | 0 | 0 | 0 | 0 | 0
  ALT OR AST > 2XULN | 0 | 0 | 0 | 0 | 0 | 0
  ANY OF ALT, AST, TOTAL BILIRUBIN OR ALP > 8XULN | 0 | 0 | 0 | 1 | 0 | 1
  TOTAL BILIRUBIN > 3XULN | 1 | 0 | 0 | 0 | 0 | 1

6. Secondary Outcome: BMS-986012 Maximum Observed Serum Concentration (Cmax)
Description: BMS-986012 maximum observed serum concentration (Cmax).
Time Frame: Cycle 1 day 1, cycle 3 day 1 (including pre-dose, 1, 2, 4, 8, 24, 72, 168, 336 hours post dose)
Population: All participants who receive at least 1 dose of BMS-986012 (and Nivolumab in the combination therapy) and have available serum concentration data for the corresponding analyte
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ug/mL
Arm/Group | BMS 70mg | BMS 160mg | BMS 400mg | BMS 1000mg | BMS 400mg + Nivo 360mg | BMS 1000mg + Nivo 360mg
Number analyzed (Participants) | 7 | 6 | 28 | 32 | 21 | 8
ug/mL
  cycle 1 day 1 | 27.5 (31) | 53.8 (28) | 121 (26) | 276 (37) | 111 (33) | 339 (25)
  cycle 3 day 1: number analyzed (Participants) | 1 | 1 | 2 | 3 | 0 | 0
  cycle 3 day 1 | 33.8 (NA) — insufficient numbers of participants | 46.9 (NA) — insufficient numbers of participants | 221 (1) | 279 (37) |  |

7. Secondary Outcome: BMS-986012 Time of Maximum Observed Serum Concentration (Tmax)
Description: BMS-986012 time of maximum observed serum concentration (Tmax).
Time Frame: Cycle 1 day 1, cycle 3 day 1 (including pre-dose, 1, 2, 4, and 8 hours post dose)
Population: as for outcome 6
Measure: Median (Full Range); unit: hours
Arm/Group | BMS 70mg | BMS 160mg | BMS 400mg | BMS 1000mg | BMS 400mg + Nivo 360mg | BMS 1000mg + Nivo 360mg
Number analyzed (Participants) | 7 | 6 | 28 | 32 | 21 | 8
hours
  cycle 1 day 1 | 2.08 [1.00 to 8.00] | 2.02 [1.00 to 6.33] | 2.00 [1.00 to 6.07] | 1.58 [0.950 to 4.40] | 4.00 [1.00 to 5.40] | 1.53 [1.00 to 4.30]
  cycle 3 day 1: number analyzed (Participants) | 1 | 1 | 2 | 3 | 0 | 0
  cycle 3 day 1 | 1.93 [1.93 to 1.93] | 4.00 [4.00 to 4.00] | 2.04 [2.02 to 2.07] | 2.30 [2.05 to 4.00] |  |

8. Secondary Outcome: BMS-986012 Area Under the Serum Concentration-time Curve From Time Zero to Time of Last Quantifiable Concentration (AUC (0-T))
Description: BMS-986012 area under the serum concentration-time curve from time zero to time of last quantifiable concentration (AUC (0-T)).
Time Frame: Cycle 1 day 1, cycle 3 day 1 (including pre-dose, 1, 2, 4, 8, 24, 72, 168, 336 hours post dose)
Population: as for outcome 6
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ug/mL
Arm/Group | BMS 70mg | BMS 160mg | BMS 400mg | BMS 1000mg | BMS 400mg + Nivo 360mg | BMS 1000mg + Nivo 360mg
Number analyzed (Participants) | 7 | 6 | 28 | 32 | 21 | 8
h*ug/mL
  cycle 1 day 1 | 3997 (31) | 5584 (55) | 18456 (32) | 36223 (40) | 16527 (31) | 45126 (24)
  cycle 3 day 1: number analyzed (Participants) | 1 | 1 | 2 | 3 | 0 | 0
  cycle 3 day 1 | 7062 (NA) — insufficient numbers of participants | 10560 (NA) — insufficient numbers of participants | 42583 (8) | 58649 (28) |  |

9. Secondary Outcome: BMS-986012 Area Under the Serum Concentration-time Curve in One Dosing Interval AUC (TAU)
Description: BMS-986012 area under the serum concentration-time curve in one dosing interval AUC (TAU).
Time Frame: Cycle 1 day 1, cycle 3 day 1 (including pre-dose, 1, 2, 4, 8, 24, 72, 168, 336 hours post dose)
Population: as for outcome 6
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ug/mL
Arm/Group | BMS 70mg | BMS 160mg | BMS 400mg | BMS 1000mg | BMS 400mg + Nivo 360mg | BMS 1000mg + Nivo 360mg
Number analyzed (Participants) | 7 | 5 | 26 | 28 | 17 | 6
h*ug/mL
  cycle 1 day 1 | 4300 (29) | 8356 (28) | 19865 (28) | 40979 (34) | 18161 (30) | 49031 (26)
  cycle 3 day 1: number analyzed (Participants) | 1 | 1 | 2 | 3 | 0 | 0
  cycle 3 day 1 | 7062 (NA) — insufficient numbers of participants | 10560 (NA) — insufficient numbers of participants | 42583 (8) | 62634 (33) |  |

10. Secondary Outcome: BMS-986012 Observed Serum Concentration at the End of a Dosing Interval (Ctau)
Description: BMS-986012 observed serum concentration at the end of a dosing interval (Ctau).
Time Frame: Cycle 1 day 1, cycle 3 day 1 (including pre-dose, 1, 2, 4, 8, 24, 72, 168, 336 hours post dose)
Population: as for outcome 6
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ug/mL
Arm/Group | BMS 70mg | BMS 160mg | BMS 400mg | BMS 1000mg | BMS 400mg + Nivo 360mg | BMS 1000mg + Nivo 360mg
Number analyzed (Participants) | 7 | 5 | 26 | 28 | 17 | 6
ug/mL
  cycle 1 day 1 | 3.44 (38) | 6.24 (31) | 17.4 (32) | 30.2 (59) | 14.6 (44) | 39.5 (40)
  cycle 3 day 1: number analyzed (Participants) | 1 | 1 | 2 | 3 | 0 | 0
  cycle 3 day 1 | 7.39 (NA) — insufficient numbers of participants | 13.6 (NA) — insufficient numbers of participants | 42.4 (13) | 59.2 (19) |  |

11. Secondary Outcome: BMS-986012 Total Body Clearance (CLT)
Description: BMS-986012 total body clearance (CLT).
Time Frame: Cycle 1 day 1, cycle 3 day 1 (including pre-dose, 1, 2, 4, 8, 24, 72, 168, 336 hours post dose)
Population: as for outcome 6
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: mL/h
Arm/Group | BMS 70mg | BMS 160mg | BMS 400mg | BMS 1000mg | BMS 400mg + Nivo 360mg | BMS 1000mg + Nivo 360mg
Number analyzed (Participants) | 7 | 5 | 26 | 28 | 17 | 6
mL/h
  cycle 1 day 1 | 16.3 (38) | 19.1 (27) | 20.1 (24) | 24.4 (86) | 22.0 (30) | 20.4 (28)
  cycle 3 day 1: number analyzed (Participants) | 1 | 1 | 2 | 3 | 0 | 0
  cycle 3 day 1 | 9.91 (NA) — insufficient numbers of participants | 15.2 (NA) — insufficient numbers of participants | 9.39 (8) | 16.0 (40) |  |

12. Secondary Outcome: BMS-986012 Trough Observed Serum Concentration (Ctrough)
Description: BMS-986012 trough observed serum concentration (Ctrough).
Time Frame: Cycle 2 day 1, cycle 3 day 1, cycle 4 day 1, cycle 7 day 1, cycle 11 day 1. cycle 15 day 1 (including pre-dose, 1, 2, 4, 8, 24, 72, 168, 336 hours post dose)
Population: as for outcome 6
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | BMS 70mg | BMS 160mg | BMS 400mg | BMS 1000mg | BMS 400mg + Nivo 360mg | BMS 1000mg + Nivo 360mg
Number analyzed (Participants) | 4 | 4 | 22 | 18 | 13 | 5
ng/mL
  cycle 2 day 1 | 4186 (27) | 7211 (17) | 18810 (29) | 36990 (54) | 14544 (84) | 36391 (43)
  cycle 3 day 1: number analyzed (Participants) | 1 | 1 | 9 | 7 | 7 | 3
  cycle 3 day 1 | 6570 (NA) — insufficient numbers of participants | 9100 (NA) — insufficient numbers of participants | 29232 (36) | 68589 (57) | 26016 (37) | 158801 (85)
  cycle 4 day 1: number analyzed (Participants) | 1 | 1 | 6 | 5 | 6 | 1
  cycle 4 day 1 | 7390 (NA) — insufficient numbers of participants | 13600 (NA) — insufficient numbers of participants | 35122 (26) | 90207 (68) | 26102 (63) | 157000 (NA) — insufficient numbers of participants
  cycle 7 day 1: number analyzed (Participants) | 1 | 1 | 4 | 4 | 3 | 0
  cycle 7 day 1 | 9040 (NA) — insufficient numbers of participants | 13700 (NA) — insufficient numbers of participants | 38315 (27) | 107444 (58) | 38405 (9) |
  cycle 11 day 1: number analyzed (Participants) | 1 | 0 | 2 | 2 | 1 | 0
  cycle 11 day 1 | 9930 (NA) — insufficient numbers of participants |  | 32251 (14) | 102980 (67) | 34400 (NA) — insufficient numbers of participants |
  cycle 15 day 1: number analyzed (Participants) | 1 | 0 | 0 | 0 | 0 | 0
  cycle 15 day 1 | 8029 (NA) — insufficient numbers of participants |  |  |  |  |

13. Secondary Outcome: BMS-986012 Average Concentration Over a Dosing Interval (Css-avg)
Description: BMS-986012 Average concentration over a dosing interval ([AUC(TAU)/tau] (Css-avg).
Time Frame: Cycle 3 day 1 (including pre-dose, 1, 2, 4, and 8 hours post dose)
Population: as for outcome 6
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ug/mL
Arm/Group | BMS 70mg | BMS 160mg | BMS 400mg | BMS 1000mg | BMS 400mg + Nivo 360mg | BMS 1000mg + Nivo 360mg
Number analyzed (Participants) | 1 | 1 | 2 | 3 | 0 | 0
ug/mL | 13.9 (NA) — insufficient numbers of participants | 22.0 (NA) — insufficient numbers of participants | 82.1 (11) | 119 (33) |  |

14. Secondary Outcome: BMS-986012 Accumulation Index (AI_AUC)
Description: BMS-986012 accumulation index. Ratio of an exposure measure at steady state to that after the first dose.
Time Frame: Cycle 3 day 1 (including pre-dose, 1, 2, 4, and 8 hours post dose)
Population: as for outcome 6
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio
Arm/Group | BMS 70mg | BMS 160mg | BMS 400mg | BMS 1000mg | BMS 400mg + Nivo 360mg | BMS 1000mg + Nivo 360mg
Number analyzed (Participants) | 1 | 1 | 2 | 2 | 0 | 0
Ratio | 1.56 (NA) — insufficient numbers of participants | 1.55 (NA) — insufficient numbers of participants | 1.62 (22) | 1.39 (51) |  |

15. Secondary Outcome: BMS-986012 Cmax Accumulation Index (AI_Cmax)
Description: BMS-986012 Cmax accumulation index (AI_Cmax). Ratio of an exposure measure at steady state to that after the first dose.
Time Frame: Cycle 3 day 1 (including pre-dose, 1, 2, 4, and 8 hours post dose)
Population: as for outcome 6
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio
Arm/Group | BMS 70mg | BMS 160mg | BMS 400mg | BMS 1000mg | BMS 400mg + Nivo 360mg | BMS 1000mg + Nivo 360mg
Number analyzed (Participants) | 1 | 1 | 2 | 2 | 0 | 0
Ratio | 0.994 (NA) — insufficient numbers of participants | 1.47 (NA) — insufficient numbers of participants | 1.22 (11) | 0.940 (70) |  |

16. Secondary Outcome: BMS-986012 Ctau Accumulation Index (AI_Ctau)
Description: BMS-986012 Ctau accumulation index (AI_Ctau). Ratio of an exposure measure at steady state to that after the first dose.
Time Frame: Cycle 3 day 1 (including pre-dose, 1, 2, 4, and 8 hours post dose)
Population: as for outcome 6
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio
Arm/Group | BMS 70mg | BMS 160mg | BMS 400mg | BMS 1000mg | BMS 400mg + Nivo 360mg | BMS 1000mg + Nivo 360mg
Number analyzed (Participants) | 1 | 1 | 2 | 2 | 0 | 0
Ratio | 1.81 (NA) — insufficient numbers of participants | 2.31 (NA) — insufficient numbers of participants | 1.76 (0) | 1.08 (82) |  |

17. Secondary Outcome: BMS-986012 Effective Elimination (T-HALFeff)
Description: BMS-986012 effective elimination (T-HALFeff) that explains the degree of accumulation observed for a specific exposure measure.
Time Frame: Cycle 3 day 1 (including pre-dose, 1, 2, 4, and 8 hours post dose)
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: Hours
Arm/Group | BMS 70mg | BMS 160mg | BMS 400mg | BMS 1000mg | BMS 400mg + Nivo 360mg | BMS 1000mg + Nivo 360mg
Number analyzed (Participants) | 1 | 1 | 2 | 1 | 0 | 0
Hours | 342 (NA) — insufficient numbers of participants | 319 (NA) — insufficient numbers of participants | 384 (154.2) | 583 (NA) — insufficient numbers of participants |  |

18. Secondary Outcome: Best Overall Response (BOR)
Description: BOR defined as the best response designation over the study as a whole. Complete Response (CR) = Disappearance of all target lesions; Partial Response (PR) = At least a 30% decrease in the sum of diameters of target lesions; Stable Disease (SD) = Neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD; Progressive Disease (PD) = At least a 20% increase in the sum of diameters of target lesions and the sum must demonstrate an absolute increase of at least 5 mm
Time Frame: From first dose to the last tumor assessment prior to subsequent therapy (Up to 97 months)
Population: All treated participants
Measure: Count of Participants; unit: Participants
Arm/Group | BMS 70mg | BMS 160mg | BMS 400mg | BMS 1000mg | BMS 400mg + Nivo 360mg | BMS 1000mg + Nivo 360mg
Number analyzed (Participants) | 7 | 6 | 29 | 35 | 21 | 8
Participants
  Complete Response | 1 | 0 | 0 | 0 | 1 | 0
  Partial Response | 0 | 0 | 1 | 1 | 8 | 2
  Stable Disease | 0 | 2 | 8 | 8 | 2 | 1
  Progressive Disease | 4 | 2 | 18 | 21 | 9 | 3
  Not evaluable | 2 | 2 | 2 | 5 | 1 | 2

19. Secondary Outcome: Objective Response Rate (ORR)
Description: ORR is defined as the percent of participants whose BOR is either CR or PR. Complete Response (CR) = Disappearance of all target lesions; Partial Response (PR) = At least a 30% decrease in the sum of diameters of target lesions; Progressive Disease (PD) = At least a 20% increase in the sum of diameters of target lesions and the sum must demonstrate an absolute increase of at least 5 mm
Time Frame: From first dose date to the date of first documented disease progression (Up to 97 months)
Population: All treated participants
Measure: Number (95% Confidence Interval); unit: Percent of participants
Arm/Group | BMS 70mg | BMS 160mg | BMS 400mg | BMS 1000mg | BMS 400mg + Nivo 360mg | BMS 1000mg + Nivo 360mg
Number analyzed (Participants) | 7 | 6 | 29 | 35 | 21 | 8
Percent of participants | 14.3 [0.4 to 57.9] | 0 [0.0 to 45.9] | 3.4 [0.1 to 17.8] | 2.9 [0.1 to 14.9] | 42.9 [21.8 to 66.0] | 25.0 [3.2 to 65.1]

20. Secondary Outcome: Duration of Response (DoR)
Description: DoR is defined as the time from first response (CR or PR) to the date of the first documented tumor progression as determined using RECIST 1.1 criteria or death due to any cause, whichever occurs first. Participants who remain alive and have not progressed will be censored on the date of their last tumor assessment.
  Complete Response (CR) = Disappearance of all target lesions; Partial Response (PR )= At least a 30% decrease in the sum of diameters of target lesions; Progressive Disease (PD) = At least a 20% increase in the sum of diameters of target lesions and the sum must demonstrate an absolute increase of at least 5 mm
  Median DOR will only be evaluated provided there are enough responding participants to warrant inclusion.
Time Frame: From the date of first dose to the date of the first documented tumor progression or death due to any cause, whichever occurs first (Up to 97 months)
Population: Median DoR is pre-specified to only be evaluated provided there are enough responders (CR or PR) to warrant inclusion (Only Cohorts with at least 5 events are analyzed)
Measure: Median (95% Confidence Interval); unit: Weeks
Arm/Group | BMS 70mg | BMS 160mg | BMS 400mg | BMS 1000mg | BMS 400mg + Nivo 360mg | BMS 1000mg + Nivo 360mg
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 9 | 0
Weeks |  |  |  |  | 120.57 [12.14 to NA] — Upper Limit not reached due to insufficient number of participants with events |

21. Secondary Outcome: Progression Free Survival (PFS)
Description: PFS is defined as the time from the date of first dose of study medication to the date of the first objective documentation of tumor progression or death due to any cause, if death occurred within 100 days after last BMS-986012 dose.
  Progressive Disease (PD) = At least a 20% increase in the sum of diameters of target lesions and the sum must demonstrate an absolute increase of at least 5 mm
Time Frame: From first dose to the date of first documented disease progression or death due to any cause, if death occurred within 100 days after last BMS-986012 dose (Up to 97 months)
Population: All treated participants
Measure: Median (95% Confidence Interval); unit: Weeks
Arm/Group | BMS 70mg | BMS 160mg | BMS 400mg | BMS 1000mg | BMS 400mg + Nivo 360mg | BMS 1000mg + Nivo 360mg
Number analyzed (Participants) | 7 | 6 | 29 | 35 | 21 | 8
Weeks | 5.50 [2.43 to 53.00] | 5.86 [5.29 to 30.29] | 5.79 [5.57 to 8.00] | 5.36 [5.00 to 5.71] | 17.71 [6.14 to 120.29] | 5.71 [2.71 to 25.00]

22. Secondary Outcome: Progression Free Survival Rate (PFSR)
Description: PFSR is defined as the percent of participants who remain progression free and surviving at "t" weeks (t= 12, 24, 36, 48, 60, 72).
  Progressive Disease (PD)=At least a 20% increase in the sum of diameters of target lesions and the sum must demonstrate an absolute increase of at least 5 mm
Time Frame: Weeks 12, 24, 36, 48, 60, 72
Population: All treated participants
Measure: Number (95% Confidence Interval); unit: Percent of participants
Arm/Group | BMS 70mg | BMS 160mg | BMS 400mg | BMS 1000mg | BMS 400mg + Nivo 360mg | BMS 1000mg + Nivo 360mg
Number analyzed (Participants) | 7 | 6 | 29 | 35 | 21 | 8
Percent of participants
  Week 12 | NA [NA to NA] — Insufficient number of participants with events | NA [NA to NA] — Insufficient number of participants with events | 21.4 [8.7 to 37.8] | 20.6 [9.1 to 35.3] | 55.0 [31.3 to 73.5] | NA [NA to NA] — Insufficient number of participants with events
  Week 24 | NA [NA to NA] — Insufficient number of participants with events | NA [NA to NA] — Insufficient number of participants with events | NA [NA to NA] — Insufficient number of participants with events | NA [NA to NA] — Insufficient number of participants with events | 45.0 [23.1 to 64.7] | NA [NA to NA] — Insufficient number of participants with events
  Week 36 | NA [NA to NA] — Insufficient number of participants with events | NA [NA to NA] — Insufficient number of participants with events | NA [NA to NA] — Insufficient number of participants with events | NA [NA to NA] — Insufficient number of participants with events | 45.0 [23.1 to 64.7] | NA [NA to NA] — Insufficient number of participants with events
  Week 48 | NA [NA to NA] — Insufficient number of participants with events | NA [NA to NA] — Insufficient number of participants with events | NA [NA to NA] — Insufficient number of participants with events | NA [NA to NA] — Insufficient number of participants with events | 35.0 [15.7 to 55.2] | NA [NA to NA] — Insufficient number of participants with events
  Week 60 | NA [NA to NA] — Insufficient number of participants with events | NA [NA to NA] — Insufficient number of participants with events | NA [NA to NA] — Insufficient number of participants with events | NA [NA to NA] — Insufficient number of participants with events | 35.0 [15.7 to 55.2] | NA [NA to NA] — Insufficient number of participants with events
  Week 72 | NA [NA to NA] — Insufficient number of participants with events | NA [NA to NA] — Insufficient number of participants with events | NA [NA to NA] — Insufficient number of participants with events | NA [NA to NA] — Insufficient number of participants with events | 35.0 [15.7 to 55.2] | NA [NA to NA] — Insufficient number of participants with events

23. Secondary Outcome: Number of Participants With Anti-BMS-986012 Antibodies (ADA)
Description: Number of participants with anti-BMS-986012 antibodies (ADA) with status as baseline ADA positive, ADA positive and ADA negative. Baseline ADA positive participant is a participant with baseline ADA positive sample (Day 1 predose). ADA-positive participant is a participant with at least one ADA positive sample relative to baseline at any time after initiation of treatment during the defined observation time period. ADA negative participant is a participant with no ADA positive sample after the initiation of treatment.
Time Frame: From first dose to 100 days following the last BMS-986012 dose (Up to 64 months)
Population: All treated participants who had at least 1 post-treatment immunogenicity assessment
Measure: Count of Participants; unit: Participants
Arm/Group | BMS 70mg | BMS 160mg | BMS 400mg | BMS 1000mg | BMS 400mg + Nivo 360mg | BMS 1000mg + Nivo 360mg
Number analyzed (Participants) | 5 | 5 | 27 | 25 | 14 | 7
Participants
  Baseline ADA positive | 0 | 0 | 0 | 1 | 0 | 0
  ADA positive | 0 | 0 | 0 | 0 | 0 | 0
  ADA negative | 5 | 5 | 27 | 25 | 14 | 7

ADVERSE EVENTS:
Time Frame: SAEs and Other AEs are assessed from first dose up to 100 days post last dose (Up to 64 months). Participants were assessed for all-cause mortality from their first dose to their study completion (Up to 97 months).
Groups:
- BMS 70mg SCLC Refractory; BMS 70mg SCLC Sensitive: 70 mg IV BMS-986012 every 21 days until protocol-specified discontinuation criteria are met
- BMS 160mg SCLC Refractory; BMS 160mg SCLC Sensitive: 160 mg IV BMS-986012 every 21 days until protocol-specified discontinuation criteria are met
- BMS 400mg SCLC Refractory; BMS 400mg SCLC Sensitive; BMS 400mg SCLC Refractory Expansion; BMS 400mg SCLC Sensitive Expansion: 400 mg IV BMS-986012 every 21 days until protocol-specified discontinuation criteria are met
- BMS 1000mg SCLC Refractory; BMS 1000mg SCLC Sensitive; BMS 1000mg SCLC Refractory Expansion; BMS 1000mg SCLC Sensitive Expansion: 1000 mg IV BMS-986012 every 21 days until protocol-specified discontinuation criteria are met
- BMS 400mg + Nivo 360mg SCLC Refractory; BMS 400mg + Nivo 360mg SCLC Sensitive; BMS 400mg + Nivo 360mg SCLC Refractory Expansion; BMS 400mg + Nivo 360mg SCLC Sensitive Expansion: 400 mg IV BMS-986012 + 360 mg Nivolumab every 21 days until protocol-specified discontinuation criteria are met
- BMS 1000mg + Nivo 360mg SCLC Refractory; BMS 1000mg + Nivo 360mg SCLC Sensitive: 1000 mg IV BMS-986012 + 360 mg Nivolumab every 21 days until protocol-specified discontinuation criteria are met
Arm/Group | BMS 70mg SCLC Refractory | BMS 70mg SCLC Sensitive | BMS 160mg SCLC Refractory | BMS 160mg SCLC Sensitive | BMS 400mg SCLC Refractory | BMS 400mg SCLC Sensitive | BMS 400mg SCLC Refractory Expansion | BMS 400mg SCLC Sensitive Expansion | BMS 1000mg SCLC Refractory | BMS 1000mg SCLC Sensitive | BMS 1000mg SCLC Refractory Expansion | BMS 1000mg SCLC Sensitive Expansion | BMS 400mg + Nivo 360mg SCLC Refractory | BMS 400mg + Nivo 360mg SCLC Sensitive | BMS 400mg + Nivo 360mg SCLC Refractory Expansion | BMS 400mg + Nivo 360mg SCLC Sensitive Expansion | BMS 1000mg + Nivo 360mg SCLC Refractory | BMS 1000mg + Nivo 360mg SCLC Sensitive
All-Cause Mortality (participants affected / at risk) | 3/3 | 4/4 | 1/2 | 1/4 | 3/3 | 3/4 | 9/12 | 9/10 | 3/3 | 5/6 | 11/12 | 12/14 | 2/2 | 6/6 | 3/4 | 4/9 | 3/3 | 5/5
Serious Adverse Events (participants affected / at risk) | 3/3 | 4/4 | 2/2 | 2/4 | 3/3 | 4/4 | 8/12 | 6/10 | 3/3 | 2/6 | 8/12 | 11/14 | 1/2 | 4/6 | 2/4 | 4/9 | 3/3 | 2/5
Other Adverse Events (participants affected / at risk) | 3/3 | 4/4 | 2/2 | 4/4 | 3/3 | 4/4 | 12/12 | 10/10 | 3/3 | 6/6 | 12/12 | 14/14 | 2/2 | 6/6 | 4/4 | 9/9 | 3/3 | 5/5
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | BMS 70mg SCLC Refractory (N=3) | BMS 70mg SCLC Sensitive (N=4) | BMS 160mg SCLC Refractory (N=2) | BMS 160mg SCLC Sensitive (N=4) | BMS 400mg SCLC Refractory (N=3) | BMS 400mg SCLC Sensitive (N=4) | BMS 400mg SCLC Refractory Expansion (N=12) | BMS 400mg SCLC Sensitive Expansion (N=10) | BMS 1000mg SCLC Refractory (N=3) | BMS 1000mg SCLC Sensitive (N=6) | BMS 1000mg SCLC Refractory Expansion (N=12) | BMS 1000mg SCLC Sensitive Expansion (N=14) | BMS 400mg + Nivo 360mg SCLC Refractory (N=2) | BMS 400mg + Nivo 360mg SCLC Sensitive (N=6) | BMS 400mg + Nivo 360mg SCLC Refractory Expansion (N=4) | BMS 400mg + Nivo 360mg SCLC Sensitive Expansion (N=9) | BMS 1000mg + Nivo 360mg SCLC Refractory (N=3) | BMS 1000mg + Nivo 360mg SCLC Sensitive (N=5)
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Cardiac tamponade (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pericardial effusion (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Adrenal insufficiency (Endocrine disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Hyperthyroidism (Endocrine disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Colitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Gastric haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Pancreatitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Retroperitoneal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Fatigue (General disorders) | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Oedema peripheral (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pain (General disorders) | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Performance status decreased (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Pyrexia (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Acute hepatic failure (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Hepatic failure (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Bacterial infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Diarrhoea infectious (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Enterocolitis infectious (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Influenza (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Lower respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0
Sepsis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Infusion related reaction (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Radiation necrosis (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Spinal fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Toxicity to various agents (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0
Hypophosphataemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pathological fracture (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 3 | 1 | 2 | 2 | 1 | 5 | 3 | 3 | 1 | 6 | 6 | 0 | 3 | 1 | 1 | 2 | 2
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cerebrovascular accident (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dysarthria (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Encephalopathy (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Transient ischaemic attack (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Confusional state (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Delirium (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Mental status changes (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Psychiatric decompensation (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Haematuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Bronchial artery hypertrophy (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Hypotension (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Superior vena cava occlusion (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | BMS 70mg SCLC Refractory (N=3) | BMS 70mg SCLC Sensitive (N=4) | BMS 160mg SCLC Refractory (N=2) | BMS 160mg SCLC Sensitive (N=4) | BMS 400mg SCLC Refractory (N=3) | BMS 400mg SCLC Sensitive (N=4) | BMS 400mg SCLC Refractory Expansion (N=12) | BMS 400mg SCLC Sensitive Expansion (N=10) | BMS 1000mg SCLC Refractory (N=3) | BMS 1000mg SCLC Sensitive (N=6) | BMS 1000mg SCLC Refractory Expansion (N=12) | BMS 1000mg SCLC Sensitive Expansion (N=14) | BMS 400mg + Nivo 360mg SCLC Refractory (N=2) | BMS 400mg + Nivo 360mg SCLC Sensitive (N=6) | BMS 400mg + Nivo 360mg SCLC Refractory Expansion (N=4) | BMS 400mg + Nivo 360mg SCLC Sensitive Expansion (N=9) | BMS 1000mg + Nivo 360mg SCLC Refractory (N=3) | BMS 1000mg + Nivo 360mg SCLC Sensitive (N=5)
Anaemia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 2 | 1 | 0 | 0 | 1 | 1 | 1 | 1 | 1 | 1 | 0 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Myelosuppression (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Atrial flutter (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Atrioventricular block second degree (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Palpitations (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Sinus tachycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Tachycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Ventricular tachycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Deafness (Ear and labyrinth disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Ear pain (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Hypoacusis (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Middle ear effusion (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vertigo (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0
Hyperthyroidism (Endocrine disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 0 | 0
Hypothyroidism (Endocrine disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 3 | 0 | 1
Cataract (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Conjunctival haemorrhage (Eye disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Diplopia (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Dry eye (Eye disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 1
Eye discharge (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Eye inflammation (Eye disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Eye irritation (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Eye pruritus (Eye disorders) | 1 | 1 | 0 | 1 | 0 | 1 | 1 | 1 | 0 | 2 | 1 | 1 | 0 | 0 | 0 | 1 | 0 | 1
Eyelid disorder (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Eyelid pain (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Eyelids pruritus (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Myopia (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Ocular hyperaemia (Eye disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Ophthalmic vein thrombosis (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Photophobia (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Retinal artery occlusion (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Swelling of eyelid (Eye disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Vision blurred (Eye disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 1
Visual impairment (Eye disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vitreous floaters (Eye disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Abdominal discomfort (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Abdominal distension (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 1 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 2 | 3 | 1 | 0 | 3 | 3 | 1 | 1 | 0 | 2 | 1 | 1
Abdominal pain lower (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 3 | 1 | 0
Aphthous ulcer (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Constipation (Gastrointestinal disorders) | 1 | 3 | 1 | 1 | 1 | 1 | 5 | 6 | 2 | 1 | 2 | 3 | 0 | 2 | 1 | 4 | 2 | 1
Defaecation urgency (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 0 | 1 | 1 | 1 | 1 | 0 | 0 | 2 | 0 | 2 | 5 | 3 | 1 | 1 | 1 | 4 | 0 | 2
Diarrhoea haemorrhagic (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Dry mouth (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 0 | 2 | 0 | 0 | 1 | 2 | 1 | 1
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 2 | 1 | 0
Dysphagia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Epigastric discomfort (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Flatulence (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Gingival pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Haemorrhoids (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Impaired gastric emptying (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Lip blister (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Mouth ulceration (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0
Nausea (Gastrointestinal disorders) | 1 | 4 | 1 | 1 | 2 | 1 | 2 | 3 | 2 | 2 | 7 | 5 | 1 | 2 | 2 | 4 | 1 | 3
Odynophagia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Oral discomfort (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Proctitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Stomatitis (Gastrointestinal disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 2 | 0 | 0 | 0 | 1 | 0 | 0
Swollen tongue (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Toothache (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 1 | 1 | 1 | 0 | 1 | 1 | 3 | 1 | 3 | 2 | 2 | 1 | 2 | 1 | 4 | 1 | 1
Asthenia (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Axillary pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Catheter site pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Chest discomfort (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 0 | 0 | 3 | 0 | 1 | 0 | 0 | 0 | 0
Chest pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 2 | 0 | 0
Chills (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 1 | 0 | 1
Face oedema (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Fatigue (General disorders) | 2 | 3 | 0 | 1 | 0 | 1 | 4 | 3 | 0 | 3 | 7 | 12 | 1 | 2 | 4 | 4 | 2 | 2
Feeling cold (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0
Gait disturbance (General disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 1 | 0 | 0 | 0
Generalised oedema (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Influenza like illness (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Infusion site erythema (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Infusion site pruritus (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Infusion site swelling (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Malaise (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 0
Mucosal dryness (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Mucosal inflammation (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Nodule (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Non-cardiac chest pain (General disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 2 | 0 | 1 | 0 | 1 | 0 | 0
Oedema (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Oedema peripheral (General disorders) | 0 | 1 | 0 | 0 | 2 | 0 | 1 | 2 | 1 | 0 | 4 | 2 | 1 | 2 | 0 | 2 | 0 | 1
Pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 1 | 2 | 0 | 1 | 0 | 1 | 0 | 1
Peripheral swelling (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Pyrexia (General disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 2
Swelling face (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Thirst (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Biliary colic (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hyperbilirubinaemia (Hepatobiliary disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Contrast media reaction (Immune system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Dust allergy (Immune system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Seasonal allergy (Immune system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Bronchitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0
Candida infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Cellulitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Conjunctivitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cystitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Diverticulitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Ear infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Escherichia pyelonephritis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Folliculitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gastroenteritis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0
Herpes virus infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hordeolum (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0
Infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Infective exacerbation of chronic obstructive airways disease (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Localised infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Lower respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0
Nail bed infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Nasopharyngitis (Infections and infestations) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 4 | 0 | 0
Oral candidiasis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 2 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Oral herpes (Infections and infestations) | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 2 | 0 | 0 | 0 | 1 | 1 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Pneumonia aspiration (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Pneumonia haemophilus (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Pustule (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0
Sinusitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 1
Skin infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Soft tissue infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Tooth abscess (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Tracheitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 1 | 1 | 0 | 2 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 1 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 3 | 0 | 0
Bone contusion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Contusion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Infusion related reaction (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 2 | 0 | 2 | 0 | 1 | 1 | 0
Post procedural urine leak (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Procedural pain (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Scratch (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Skin abrasion (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Wound (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Alanine aminotransferase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 1 | 0 | 0
Amylase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 1
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 2 | 0 | 0
Bacterial test positive (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Blood alkaline phosphatase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Blood bilirubin increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Blood creatinine increased (Investigations) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 1 | 1 | 0 | 0
Body temperature fluctuation (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Body temperature increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Clostridium test positive (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Electrocardiogram QT prolonged (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Gamma-glutamyltransferase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
General physical condition abnormal (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
International normalised ratio increased (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Lipase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 1
Platelet count decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Staphylococcus test positive (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Streptococcus test positive (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Vitamin D decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Weight decreased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 1 | 3 | 2 | 0 | 0 | 1 | 1 | 1 | 0
Weight increased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
White blood cell count decreased (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 2 | 1 | 1 | 1 | 1 | 2 | 6 | 7 | 1 | 2 | 5 | 6 | 0 | 2 | 2 | 1 | 2 | 1
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 0 | 0 | 1 | 0
Fluid retention (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0
Glucose tolerance impaired (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 0 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Hypernatraemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 1 | 1 | 0 | 2 | 1 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 2 | 0 | 2
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 3 | 2 | 0 | 0 | 0 | 4 | 0 | 1 | 0 | 0 | 3 | 0 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 0 | 2 | 0 | 1 | 1 | 1 | 1 | 0 | 2
Hypophagia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypophosphataemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 | 1 | 0 | 1 | 0 | 1 | 3 | 1 | 0 | 0 | 2 | 1 | 1 | 2 | 2 | 9 | 1 | 3
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1 | 1 | 2 | 0 | 1 | 4 | 0 | 2 | 4 | 2 | 2 | 3 | 1 | 3 | 0 | 2
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Bursitis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Groin pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Muscle twitching (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 2 | 2 | 0 | 0 | 0 | 1 | 1 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 1 | 1 | 1 | 0 | 1 | 0 | 2 | 0 | 0
Musculoskeletal disorder (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 1 | 0 | 2 | 1 | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 0 | 0 | 1 | 0 | 2
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 1 | 0 | 1 | 1 | 2 | 0 | 1 | 3 | 1 | 0 | 0 | 1 | 2 | 0 | 2
Pain in jaw (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Pathological fracture (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Polymyalgia rheumatica (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Synovial cyst (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Tendon pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Ataxia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Balance disorder (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Burning sensation (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Cerebral ischaemia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Cerebrovascular accident (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cognitive disorder (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dementia Alzheimer's type (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Depressed level of consciousness (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Disturbance in attention (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 2 | 1 | 0 | 1 | 0 | 0 | 0 | 2 | 0 | 1 | 0 | 1 | 0 | 2 | 1 | 1 | 0 | 1
Dysaesthesia (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dysarthria (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dysgeusia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0
Dysmetria (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Headache (Nervous system disorders) | 0 | 2 | 0 | 1 | 0 | 2 | 0 | 1 | 1 | 0 | 2 | 1 | 2 | 2 | 1 | 0 | 1 | 2
Hemiparesis (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypersomnia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Hypoaesthesia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 1
Memory impairment (Nervous system disorders) | 0 | 1 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 0
Myoclonus (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Neuralgia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Neuropathy peripheral (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0
Paraesthesia (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 2 | 1 | 1 | 0 | 1 | 2 | 0 | 1
Parosmia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Peripheral sensory neuropathy (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 2 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 2 | 0 | 0
Peroneal nerve palsy (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Presyncope (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Restless legs syndrome (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Somnolence (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Syncope (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Transient ischaemic attack (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Tremor (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Abnormal dreams (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Agitation (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Anxiety (Psychiatric disorders) | 0 | 2 | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 1
Confusional state (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 2 | 1 | 0 | 1 | 0 | 0 | 1
Delirium (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Depression (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Disorientation (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hallucination (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Insomnia (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 3 | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 3 | 1 | 0
Mood altered (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Restlessness (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Acute kidney injury (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0
Dysuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Haematuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Hydronephrosis (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Leukocyturia (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Nocturia (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0
Pollakiuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Proteinuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Renal disorder (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Renal failure (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Urinary incontinence (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Urinary tract pain (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Acquired phimosis (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Genital burning sensation (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pelvic pain (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Penile erythema (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Pruritus genital (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Vulvovaginal burning sensation (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Vulvovaginal pruritus (Reproductive system and breast disorders) | 1 | 2 | 1 | 1 | 0 | 0 | 0 | 1 | 0 | 2 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 2
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0 | 1 | 1 | 1 | 1 | 1 | 0 | 2 | 0 | 3 | 1 | 0 | 1 | 4 | 0 | 0
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 1 | 1 | 0 | 2 | 1 | 2 | 1 | 2 | 2 | 0 | 0 | 0 | 3 | 1 | 1
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 1 | 0 | 0 | 0 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Laryngeal haemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Nasal dryness (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 3 | 0 | 2 | 0 | 2 | 0 | 2
Pulmonary haemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Rales (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 1
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Sneezing (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 3 | 1 | 0 | 0 | 0 | 0 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 3 | 0 | 0
Dermal cyst (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 1 | 0 | 1 | 1 | 3 | 1 | 3
Eczema (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0
Erythema (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 1
Erythema multiforme (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Hand dermatitis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Miliaria (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Nail disorder (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Nail hypertrophy (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Night sweats (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Onychoclasis (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Onychomadesis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Pain of skin (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Palmar erythema (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Pemphigoid (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Petechiae (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 0 | 0
Photosensitivity reaction (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 2 | 4 | 2 | 2 | 3 | 4 | 12 | 8 | 3 | 6 | 9 | 13 | 1 | 5 | 4 | 9 | 3 | 5
Psoriasis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Purpura (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 2 | 0 | 0 | 0 | 2 | 0 | 2 | 0 | 0 | 0 | 0
Rash erythematous (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Rash macular (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 3 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Rash papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Rash pruritic (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Rash vesicular (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 1
Scab (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Skin discolouration (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Skin disorder (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Skin exfoliation (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Skin lesion (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 1
Skin mass (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Deep vein thrombosis (Vascular disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Embolism (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Flushing (Vascular disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0
Hot flush (Vascular disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypertension (Vascular disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Hypotension (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Poor venous access (Vascular disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Bristol-Myers Squibb Co. agreements with investigators vary; constant is our right to embargo communications regarding trial results prior to public release for a period ≤60 days from submittal for review. We will not prohibit investigators from publishing but will prohibit the disclosure of previously undisclosed confidential information other than study results, and request postponement of single-center publications until after disclosure of the clinical trial's primary publication.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-06-06): https://cdn.clinicaltrials.gov/large-docs/49/NCT02247349/Prot_SAP_000.pdf